CLINICAL TRIAL: NCT02744300
Title: Diabetes Prevention in Women With a Recent History of Gestational Diabetes Mellitus
Brief Title: Balance After Baby Intervention for Women With Recent Gestational Diabetes
Acronym: BABI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Ellen W. Seely, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6201.25-S01
Record Dates: First submitted 2016-03-03; First posted 2016-04-20 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus (GDM) in most recent pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BABI-2 Lifestyle Intervention (Experimental): Participants in this group will take part in the web-based lifestyle intervention which includes access to the lifestyle intervention website and personalized coaching from a Lifestyle Coach.
  Interventions: Behavioral: BABI-2 Lifestyle Intervention
- Post-GDM Follow-up Group (No Intervention): Participants in this group will have access to a separate website containing links to information about diabetes prevention.

INTERVENTIONS:
Behavioral: BABI-2 Lifestyle Intervention — Participants in this intervention will receive support from a lifestyle coach and gain access to a website with online presentations that contain healthy eating and physical activity educational tips.
  Other Names: Balance After Baby 2 Lifestyle Intervention Program
  Arms: BABI-2 Lifestyle Intervention

SUMMARY:
Women with a history of gestational diabetes mellitus (GDM) have an increased risk of developing type 2 diabetes later in life. In our 2012 pilot study we created and tested a web-based lifestyle intervention program adapted from the NIH sponsored Diabetes Prevention Program (DPP), modified specifically for women with a recent history of GDM. This program, delivered in the first year postpartum, encouraged weight loss, dietary changes, and physical activity. The purpose of the current study, called Balance After Baby Intervention 2 (BABI-2), is to study a larger group of women with two years of follow-up. We will assess whether women assigned to the intervention group lose more weight and decrease their risk factors for type 2 diabetes.

Participants assigned to the BAB lifestyle intervention will receive support from a lifestyle coach and gain access to a website with online presentations that contain healthy eating and physical activity educational tips.

Participants assigned to the post-GDM follow-up group will have access to a website containing links to information about diabetes prevention.

DETAILED DESCRIPTION:
The landmark Diabetes Prevention Program (DPP) demonstrated that an intensive lifestyle intervention in people with impaired glucose tolerance (IGT) could reduce the incidence of type 2 diabetes. These findings were consistent, regardless of ethnicity, age, body mass index (BMI), gender. However, the DPP does not have a specific focus on new mothers with a recent history of gestational diabetes. Although there are recommendations that all women with gestational diabetes mellitus (GDM) receive postpartum testing for diabetes and type 2 diabetes risk reduction, study findings suggest that women with a recent history of GDM may be unaware of their risk for future diabetes, and also do not take steps to reduce their risks.

The postpartum period is also a time when many changes occur in a woman's life, with competing responsibilities often altering sleep patterns, work schedules, eating patterns, exercise regularity, and time allocation. New mothers may have difficulty engaging in healthy lifestyle programs because of lack of time and energy, and because of competing work and family demands, including child care. In response to the barriers identified in literature and gleaned from the focus groups and informant interviews of a preliminary study (2009p000042), we created a lifestyle/behavioral intervention that utilizes a modified DPP.

In 2012 we completed a one year pilot study (2009p002118) to assess the feasibility and effectiveness of the lifestyle/behavioral intervention. The pilot study demonstrated that women in the intervention group lost more weight and were closer to pre-pregnancy weight that the control group.

Our goals in Phase 2 of the study are: to gather more data about the effects of the intervention at 12 months; to determine if the greater weight loss observed in the pilot intervention arm at 12 months can be replicated with a larger number of women and maintained at 24 months; and to see whether there is a significant effect on glucose tolerance in the intervention arm at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female with a diagnosis of gestational diabetes mellitus (GDM) by Carpenter-Coustan criteria (see below) in most recent singleton or twin pregnancy (Carpenter & Coustan, 1982)
* Women with a glucose value ≥200 mg/dL after a 50-g glucose challenge test at >12 weeks' gestation will also be included
* 18 years of age or older
* No personal history of Type 1 or 2 diabetes
* Pre-pregnancy body mass index between 18 and 50 kg/m2
* Six weeks postpartum body mass index between 24 and 50 kg/m2 (>22 for Asians)
* Daily access to the internet
* English or Spanish speaking
* Capable of providing informed consent

Exclusion Criteria:

* Pre-pregnancy diagnosis of diabetes (type 1, 2, or a secondary form of diabetes)
* Current pregnancy
* Premature delivery < 34 weeks gestation
* Diagnosis of diseases associated with glucose metabolism
* Current or planned participation in a commercial weight loss program (i.e. Jenny Craig) over the duration of the study
* Taking certain prescription medications including high dose glucocorticoids, atypical antipsychotics associated with weight gain (such as risperdal (risperidone), clozapine (clozaril), olanzapine (zyprexa), quetiapine (seroquel), etc.), or other prescription weight loss medications
* Personal history of breast cancer or any other type of cancer other than a basal cell skin cancer
* Personal history of cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication), kidney disease, liver disease, venous or arterial thromboembolic disease, adrenal insufficiency, depression requiring hospitalization within the past 6 months, or non-pregnancy related illness requiring overnight hospitalization in the past 6 months
* Underlying disease/treatment that might interfere with participation in/completion of the study (e.g., significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)
* Other active medical problems detected by examination or laboratory testing
* Plans to be in a different geographic area within the next 6 months
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months after delivery
  Postpartum weight loss will be measured from 6 weeks postpartum to 12 months postpartum.

SECONDARY OUTCOMES:
Weight loss | 24 months after delivery
  Postpartum weight loss will be measured from 6 weeks postpartum to 24 months postpartum
Diabetes | 6 weeks, 12 months, and 24 months after delivery
  Risk factors or diagnosis of diabetes will be assessed in all participants via oral glucose tolerance tests (OGTTs) and by measuring glycated hemoglobin (HbA1c).
Number of participants with a fasting glucose level greater than 100 mg/dL | 6 months and 18 months postpartum
Number of participants with either: a HbA1c value greater than or equal to 5.7; or a 2 hour value on a 75 g oral glucose tolerance test of greater than or equal to 140 | 6 weeks, 12 months, and 24 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Seely, MD, Principal Investigator — Brigham and Women's Hospital; Jacinda Nicklas, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Kim SY, England L, Wilson HG, Bish C, Satten GA, Dietz P. Percentage of gestational diabetes mellitus attributable to overweight and obesity. Am J Public Health. 2010 Jun;100(6):1047-52. doi: 10.2105/AJPH.2009.172890. Epub 2010 Apr 15. PMID 20395581
- [Background] Swan W, Kilmartin G, Liaw ST. Assessment of readiness to prevent type 2 diabetes in a population of rural women with a history of gestational diabetes. Rural Remote Health. 2007 Oct-Dec;7(4):802. Epub 2007 Nov 19. PMID 18020897
- [Background] Walker LO, Grobe SJ. The construct of thriving in pregnancy and postpartum. Nurs Sci Q. 1999 Apr;12(2):151-7. doi: 10.1177/089431849901200216. PMID 11847682
- [Background] Nicklas JM, Zera CA, England LJ, Rosner BA, Horton E, Levkoff SE, Seely EW. A web-based lifestyle intervention for women with recent gestational diabetes mellitus: a randomized controlled trial. Obstet Gynecol. 2014 Sep;124(3):563-570. doi: 10.1097/AOG.0000000000000420. PMID 25162257
- [Derived] Rosenberg EA, Seely EW, James K, Soffer MD, Nelson S, Nicklas JM, Powe CE. Carbohydrate Intake and Oral Glucose Tolerance Test Results in the Postpartum Period. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1007-e1012. doi: 10.1210/clinem/dgad234. PMID 37097924